CLINICAL TRIAL: NCT03179267
Title: Detection of Physiological Deterioration by the SNAP40 Wearable Device Compared to Standard Monitoring Devices in the Emergency Department
Brief Title: Detection of Deterioration by SNAP40 Versus Standard Monitoring in the ED
Acronym: SNAP40ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Collaborators: SNAP40 (Unknown); University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/SS/0028
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2017-04

CONDITIONS: Vital Signs
Keywords: vital signs; monitoring; early warning score

STUDY DESIGN:
Intervention Model Description: Addition to standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SNAP40 monitor (Experimental): All participants in the study will be fitted with the SNAP40 ambulatory monitoring device as well as usual monitoring as standard care
  Interventions: Device: SNAP40

INTERVENTIONS:
Device: SNAP40 — SNAP40 ambulatory monitoring device

SUMMARY:
In recent years there has been increasing focus on the earlier detection of deterioration in the clinical condition of hospital patients with the aim of instigating earlier treatment to reverse this deterioration and prevent adverse outcomes. This is especially important in the ED, a dynamic environment with large volumes of undifferentiated patients, which carries inherent patient risk. SNAP40 is an innovative medical-grade device that can be worn on the upper arm that continuously monitors patients' vital signs including relative changes in systolic blood pressure, respiratory rate, heart rate, movement, blood oxygen saturation and temperature. It uses automated risk analysis to potentially allow clinical staff to easily and quickly identify high-risk patients. The aim of this study is to investigate whether the SNAP40 device is able to identify deterioration in the vital sign physiology of an ED patient earlier than current standard monitoring and observation charting techniques.

DETAILED DESCRIPTION:
As well as the potential of the SNAP40 device to improve patient safety, we believe that the SNAP40 device will increase ED efficiency, improve and increase use of resources and enable improved patient flow through the ED. Currently the only option for continuous monitoring or regular observations in the ED is to connect the patient to a standard monitor. Whilst these monitors can be portable they are not lightweight enough to allow the patient to be ambulatory within the ED and therefore require the patient to have a bed and a bed space or cubicle. This leads to lack of space within the ED, less cubicles (which allow privacy) free for performing history taking, examination and procedures, difficulty accessing patients and difficulty transporting them to areas where specialist tests can be performed (i.e. radiology and ECG). SNAP40 may remove the need for patients to be confined to beds and bed spaces (unless clinically required) freeing up space within the ED and allowing the ED care processes to occur much more freely increasing efficiency and speed of patient processing. This will undoubtedly lead to improved patient experiences around their ED and hospital journey.

The SNAP40 device also has the potential to free up resources, which can be used to improve patient care and experience in the ED. SNAP40 may reduce clinical staff time taken to record observations enabling them to provide patients with other aspects of care (i.e. analgesia and treatments) more regularly and in a timelier manner. Clinical staff may be able to spend more time with patients allowing better quality communication with them and their relatives. There will potentially be more time for traditional nursing care and personal care.

Whilst there are some other similar medical devices on the market (i.e. www.biovotion.com, www.sensium-healthcare.com, www.vitalconnect.com, http://www.caretakermedical.net) using wristbands, patches or finger cuff technology, currently none are being used in ED clinical practice.

This study will examine the SNAP40 device by comparing its performance to detect physiological deterioration against standard observations taken by clinical staff (nurses, doctors and clinical support workers) within the ED. The study will assess whether the device is able to detect physiological derangement sooner that standard monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

1. Participant aged 16 years or over AND
2. Participant triaged to Majors (High Dependency or Immediate Care) OR Participants who are stepped down from Resuscitation room care to High Dependency or Immediate Care

Exclusion Criteria:

1. Participants under 16 years of age
2. Previous participation in the study
3. Participant in custody
4. Participants deemed high risk for absconding by clinical staff
5. Participants unable to communicate in English
6. Participants who are triaged to immediate resuscitation. These participants may be considered for inclusion once immediate assessment and treatment have been initiated and they are stepped down to High Dependency (HD)/Immediate Care (IC) areas
7. Patients with implantable defibrillators, pacemakers or neurostimulators will be excluded
8. Patients who cannot have blood pressure measured in both arms e.g. patients with renal fistula, a Peripherally Inserted Central Catheter (PICC) line or who have had a lymph node clearance

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Time to detection of deterioration | 4 hours
  Time to detection of deterioration in an ED patient's vital sign physiology defined as an increase in NEWS score. This would include a deterioration in blood pressure, pulse/heart rate, respiratory rate, skin temperature (SNAP40)/core temperature (Standard), oxygen saturation reading or movement (SNAP40)/GCS (Standard).

SECONDARY OUTCOMES:
Staff observation and responding to alarm times | 4 hours
  Time ED staff spend performing a charting observations and responding to standard monitoring alarms.
Percentage clinical escalation of care when deterioration detected. | 4 hours
  Percentage clinical escalation of care when deterioration detected.
Participants satisfaction | 4 hours
  Participants rating of experience of both SNAP40 and current monitoring.
Staff satisfaction | 4 hours
  ED staff rating of experience of both SNAP40 and current monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Reed, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reed MJ, McGrath M, Black PL, Lewis S, McCann C, Whiting S, O'Brien R, Grant A, Harrison B, Skyrme L, Odam M. Detection of physiological deterioration by the SNAP40 wearable device compared to standard monitoring devices in the emergency department: the SNAP40-ED study. Diagn Progn Res. 2018 Sep 3;2:18. doi: 10.1186/s41512-018-0040-7. eCollection 2018. PMID 31093566